CLINICAL TRIAL: NCT06390566
Title: Evolution of the Functional and Muscular State and Quality of Life of Patients With Limb-girdle Muscular Dystrophy 2A: CALNATHIS Prospective Cohort Study
Brief Title: Evolution of the Functional and Muscular State of Patients With Muscular Dystrophy 2A Belts
Acronym: CALNATHIS
Status: Active, not recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230610
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Limb Girdle Muscular Dystrophy
Keywords: LGMD2A; NSAD; ACTIVLIM; 10MWT; MRI
MeSH Terms: conditions — Muscular Dystrophies, Limb-Girdle; Limb-girdle muscular dystrophy type 2A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — During the V1 inclusion visit, the information leaflet will be given to the patient, the inclusion and non-inclusion criteria will be checked and the patient will sign the consent form.
  On the morning of the 1st day of the V1 inclusion visit, demographic data/medical history/diseases will be collected. A physical examination including taking vital signs, grading according to the Brooke and Vignos scales and MRC muscle testing will be carried out. Following this, samples for the biobank (hematology, biochemistry and coagulation) will be taken.
  In the afternoon, a muscular MRI/MRS will be performed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: calpaïnopathies — Identify and quantify the loss of strength of upper and lower limb muscle groups in patients with LGMD2A
  Other Names: LGMD2A

SUMMARY:
Limb girdle muscular dystrophies were originally defined as a postnatal progressive muscle disease, which begins and primarily affects the pelvic and scapular muscles.

DETAILED DESCRIPTION:
Intro:

Limb girdle muscular dystrophies were originally defined as a postnatal progressive muscle disease, which begins and primarily affects the pelvic and scapular muscles.

To be considered a form of limb-girdle muscular dystrophy, according to the European Neuromuscular Center, the condition must be described in at least two unrelated families with affected individuals achieving independent walking, must have elevated serum creatine kinase activity, must demonstrate degenerative changes on muscle imagery over the course of the disease, and must exhibit dystrophic changes on muscle histology, ultimately leading to end-stage pathology for the most affected muscles.

They are classified into dominant forms (LGMD 1, old nomenclature; LGMD D, new nomenclature) and recessive forms (LGMD 2, old nomenclature; LGMD R new nomenclature). Recessive forms predominate in terms of number of subtypes and individual prevalence, with regional variations due to founder effects in some cases (Murphy et al, 2015).

Individually, distinct subtypes of LGMD are relatively rare; however, as a group, the minimum prevalence of LGMD is probably between 2.27 per 100,000 and 10 per 100,000. In Europe and the United States, calpainopathies, also called LGMD R1 or LGMD-2A (OMIM 253600 ), are the most common of the different types of LGMD, accounting for up to 30% of all cases of recessive LGMD.

There is currently no cure for the disease, the management of which is still based on rehabilitation therapies and the prevention of other complications. The development of new therapeutic approaches, in particular gene therapies, requires the best possible characterization of the natural history of the disease, in order to identify the patients with the most unfavorable evolutions and to characterize their chronology, and in order to identify the clinical and paraclinical parameters that are most sensitive to change, allowing the effectiveness of new treatments to be better assessed in future randomized trials. However, there are currently no or few recent data from prospective cohorts representative of the population of interest and including detailed phenotyping data such as muscle MRI.

Hypothesis/Objective

Primary objective :

The main objective of this study is to identify and quantify the loss of strength of the muscle groups of the upper (e.g.: raising the arms, lifting a weight, etc.) and lower (e.g.: walking, standing, etc.) limbs over a period of time. of 2 years in 25 patients suffering from LGMD2A already followed at the Reference Center for Neuromuscular Diseases of Mondor Hospital.

Secondary objectives:

* Define the evaluation criteria (scales, measurements) capable of defining the therapeutic response after the gene therapy clinical trial,
* Describe the loss of muscle functions (inability to raise the arms, wheelchair) and muscle weakness of the upper and lower limbs,
* Identify and monitor imaging and laboratory analysis parameters which are indicators of the progression of the disease leading to muscle deficit.

Method

Primary evaluation criteria:

Assessment of motor function • Assessment of change from baseline in motor function assessed with the North Star Assessment (NSAD) scale score for Limb Girdle Muscular Dystrophies.

Secondary evaluation criteria:

Assessment of motor function of the upper and lower limbs

* Assessment of motor function of the upper and lower limbs with the Brooke and Vignos scales Assessment of muscle strength
* 1) Isometric manual muscular assessment
* 2) Quantitative isometric muscle evaluations (Quantitative Muscle Testing (QMT))

  - Myotools and manual dynamometer (Hand Held Dynamometry (HHD)) Assessment of motor function of the upper limbs
* Assessment of the upper limbs using the PUL (Performance of the Upper Limb) assessment tool, filmed version using 3 cameras Assessment of movement activity Walking Ability Using the FeetMe® Monitor Muscle MRI
* Muscle anatomy (volume, fatty infiltration)
* Modified Mercuri Score (mMS) to measure fat splitting Laboratory analysis

Biobank samples:

* Blood sampling for hematology analyzes
* Blood sampling for biochemistry analysis (CK)
* Blood sampling for coagulation analysis Quality of life questionnaire
* Quality of life questionnaire for genetic neuromuscular diseases (gNMD) and ACTIVLIM questionnaire

Conclusion The overall objective of the analyzes planned in this study is to characterize disease progression in patients with LGMD2A over a period of up to 24 months. The choice of a study duration of 24 months is linked to the fact that over a shorter period significant changes would not have been observable and a longer duration would have greatly increased the burden and scale of the study at the time. logistical level. It is important to develop detailed natural history data to better understand the driving course of the disease and validate assays as well as clinical outcome measures to define relevant endpoints for future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of autosomal recessive LGMD2A (two pathogenic mutations in the calpain 3 gene)
* Ability to participate in the tests and examinations planned by the study (manual muscle tests, motor scales)
* Informed and having signed a consent form
* Affiliate to a social security scheme in France (beneficiary or entitled person).

Exclusion Criteria:

* Patient with another disease likely to significantly interfere with the interpretation of the natural history of LGMD2A
* Participant in a clinical trial with an investigational product within 3 months preceding inclusion
* Patient unable or unwilling to comply with protocol requirements
* Patient under guardianship, curatorship or legal protection
* Pregnant or breastfeeding woman
* Patient deprived of liberty
* Adult patient unable to express consent
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with LGMD2A already followed at the Reference Center for Neuromuscular Diseases at Henri Mondor Hospital
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2027-05-28 (Estimated); Study Completion 2027-05-28 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the loss of strength of muscle groups in patients with LGMD2A | 2 years
  identify and quantify the loss of strength of upper and lower limb muscle groups in patients with LGMD2A

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Henri Mondor, Créteil, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided